CLINICAL TRIAL: NCT01713517
Title: Impact of Insecticide Resistance in Anopheles Arabiensis on the Effectiveness of Malaria Vector Control in Sudan
Brief Title: Impact of Insecticide Resistance on Vector Control
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Federal Ministry of Health, Sudan (Other Government); World Health Organization (Other); Liverpool School of Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WHO_IR_SUDAN
Record Dates: First submitted 2012-10-22; First posted 2012-10-24 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Malaria, Falciparum
Keywords: Mosquito Control; Insecticide Resistance
MeSH Terms: conditions — Malaria, Falciparum | interventions — Pesticides; bendiocarb; decamethrin; Insecticide-Treated Bednets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Universal coverage of Long Lasting Insecticidal Nets (LLIN) (Active Comparator): Distribution of long lasting insecticidal nets to all community members in the study arm allowing for at least one net per 2 persons
  Interventions: Device: Long Lasting Insecticidal Nets (LLIN)
- LLIN Plus Indoor Residual Spraying (Experimental): Distribution of long lasting insecticidal nets to all community members in the study arm allowing for at least one net per 2 persons plus indoor residual spraying with insecticide of interior walls of all houses twice yearly.
  Interventions: Other: Indoor residual insecticide spraying (IRS); Device: Long Lasting Insecticidal Nets (LLIN)

INTERVENTIONS:
Other: Indoor residual insecticide spraying (IRS) — Application of insecticide to interior walls of domiciliary structures to kill malaria vector mosquitoes which rest on walls after taking human blood meal
  Other Names: IRS; Pesticide; Bendiocarb; Deltamethrin
  Arms: LLIN Plus Indoor Residual Spraying
Device: Long Lasting Insecticidal Nets (LLIN) — Provision of LLIN to all community members in the clusters allocated to the study arm. LLIN protect individuals from bites by malaria vector mosquitoes by providing a physical barrier and insecticidal and repellent effect.
  Other Names: Insecticide Treated Nets (ITN); Permanet2.0

SUMMARY:
The purpose of the study is to determine whether long lasting insecticidal nets and indoor residual insecticide spraying, alone or in combination, are effective for controlling insecticide resistant anopheles mosquitoes for malaria prevention.

DETAILED DESCRIPTION:
The study will assess the impact that insecticide resistance has on the effectiveness of malaria vector control tools LLIN and IRS. This is done by a cluster randomised trials of universal coverage LLINs versus universal coverage LLINs in combination with IRS, with levels of baseline insecticide resistance in the main vector balanced between the two study arms. In each cluster resistance to the insecticide used on LLINs is monitored, and malaria incidence is estimated from cluster specific cohorts of children followed up over the duration of the study. Resistance impact will be assessed from the ratio of incidence rates in clusters with high compared to those with low resistance and from a continuous measure of resistance expressed as percentage loss of mosquito mortality when exposed to insecticide in standardised WHO tests. Resistance mechanisms will be studied in subsets of study clusters.

ELIGIBILITY:
Inclusion Criteria:

* Children older than 6 months and younger than 10 years in approximately 100 randomly selected households in all 140 study clusters selected in the four study areas

Exclusion Criteria:

* Children living in households within 1 km from the edge of a neighbouring cluster (the buffer zone)

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28000 (Estimated)
Dates: Start 2011-04; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Malaria Incidence | 3 years
  Infection with malarial parasites determined by rapid diagnostic tests/microscopy in cohort members who report or have fever (>37.5C)

SECONDARY OUTCOMES:
Prevalence of P.falciparum Infection | 3 years
  Infection with plasmodial parasites (falciparum and/or vivax) in randomly selected members of the study cohort in each study cluster during the peak of the malaria transmission season by rapid diagnostic test
Entomological Innoculation rate | Average for months Sept, Oct, Nov for years 2011, 2012, 2013
  Anopheles arabiensis mosquitoes collected in sentinel clusters by light trap, window trap, clay pot and pyrethrum sheet collection and determination of sporozoite, human blood index, feeding and resting behaviour.
Frequency of insecticide resistance associated genotypes (kdr) in anopheles arabiensis | Yearly average 2011, 2012, 2013, 2014
  Molecular analysis of mosquito specimens caught in subset of clusters by pyrethrum spray collection.

CONTACTS AND LOCATIONS:
Overall Officials: Immo Kleinschmidt, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Martin J Donnelly, PhD, Principal Investigator — Liverpool School of Tropical Medicine; Khalid A Elmardi, MD, Study Director — Federal Ministry of Health, Sudan; Hmooda T Kafy, MSc, Principal Investigator — Federal Ministry of Health, Sudan; Bashir A Ismail, MSc, Principal Investigator — Federal Ministry of Health, Sudan; Mohamed Ahmed A Mohamed, MSc, Principal Investigator — Federal Ministry of Health, Sudan
Locations (3):
- Sudan (3):
  - Malaria Control Programme, Wad Medani, Al Jazirah
  - Malaria Control Programme, Gedarif, Gedarif State
  - Malaria Control Programme, Kassala, Kassala

REFERENCES:
- [Derived] Kafy HT, Ismail BA, Mnzava AP, Lines J, Abdin MSE, Eltaher JS, Banaga AO, West P, Bradley J, Cook J, Thomas B, Subramaniam K, Hemingway J, Knox TB, Malik EM, Yukich JO, Donnelly MJ, Kleinschmidt I. Impact of insecticide resistance in Anopheles arabiensis on malaria incidence and prevalence in Sudan and the costs of mitigation. Proc Natl Acad Sci U S A. 2017 Dec 26;114(52):E11267-E11275. doi: 10.1073/pnas.1713814114. Epub 2017 Dec 11. PMID 29229808